CLINICAL TRIAL: NCT06214962
Title: Comprehensive Dementia Management : From Translational Medicine to Innovative Care--Innovative Care Model for Community Care Center and Day-Care Center: Development of Classification Standard for Precision Care
Brief Title: Comprehensive Dementia Management : From Translational Medicine to Innovative Care
Status: Recruiting | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-SV(I)-20220016
Record Dates: First submitted 2023-03-13; First posted 2024-01-22 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-03

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — myotubularin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: (multiple training modalities, MTM) — 1. Invite experts to discuss the course content of each unit of MTM, and then invite teachers to take pictures , and combine them into one course for the benefit of the elderly in the institution.
  2. Select 3 units to try out in the dementia base, and make corrections based on the feedback of the elders and the base staff.
  3. Continue to complete other units based on the experience of the first 3 units.
  (2) In the Rizhao part, experts are mainly used to develop various course modules suitable for the elderly with dementia in Rizhao, and each module unit is tested on the elderly with dementia and then revised The planning task is mainly to establish a solution strategy. The method is to set up an "activity course module planning or design group" to develop various course modules suitable for Rizhao demented elders.

SUMMARY:
The purpose of this stage is to conduct analysis and discussion through expert meetings (consultation) based on the current data of the elderly in each dementia base and Rizhao Center, as well as the weekly courses and activities of the service site (base, Rizhao), and make recommendations.

DETAILED DESCRIPTION:
(1) Course content confirmation: (A) Continuing the results of the first-stage expert meeting, experts in various fields will be divided into groups to form an "activity curriculum planning group" (such as humanities and society, psychology, medical personnel, family members of dementia, etc.), and based on empirical research (type, Time, frequency, etc.) as a planning basis to develop care plans for different types of community dementia service locations and verify their effectiveness.

According to empirical research, such as for different types (dementia or mixed type) of strongholds or sunshine, plan compulsory (common activity) courses, and plan elective activity courses according to different attributes or needs, such as:

1. Common compulsory activities: physical fitness exercise, cognitive training, physical fitness combined with cognition, etc., and plan the dosage (intensity, each time and weekly frequency, etc.) according to the low, medium and high differences in physical fitness;
2. Elective activity courses: Considering the elder attributes of each service location to plan "group common elective" and "individual elective" activities, such as: integrating favorite music elements and nostalgic elements of personal life experience into "daily life activities" The main activities (such as: planting/gardening, cooking, shopping or going out, etc.

(B) Solicit and establish a connection and cooperation model between the community service organization and surrounding resources (such as clinics, foundations, volunteer groups, universities, etc.) Jointly participate in the care plan of this service agency.

The research team develops modular courses and establishes a professional teacher group for each module to provide teaching materials for service locations and personnel training.

(A) Continuing the results of the first-stage expert meeting, experts in various fields will be divided into groups to form an "activity curriculum planning group" (such as humanities and society, psychology, medical personnel, family members of dementia, etc.), and based on empirical research (type, Time, frequency, etc.) as a planning basis to develop care plans for different types of community dementia service locations and verify their effectiveness.

According to empirical research, such as for different types (dementia or mixed type) of strongholds or sunshine, plan compulsory (common activity) courses, and plan elective activity courses according to different attributes or needs, such as:

1. Common compulsory activities: physical fitness exercise, cognitive training, physical fitness combined with cognition, etc., and plan the dosage (intensity, each time and weekly frequency, etc.) according to the low, medium and high differences in physical fitness;
2. Elective activity courses: Considering the elder attributes of each service location to plan "group common elective" and "individual elective" activities, such as: integrating favorite music elements and nostalgic elements of personal life experience into "daily life activities" The main activities (such as: planting/gardening, cooking, shopping or going out, etc.

(B) Solicit and establish a connection and cooperation model between the community service organization and surrounding resources (such as clinics, foundations, volunteer groups, universities, etc.) Jointly participate in the care plan of this service agency.

(C) The research team develops modular courses and establishes a professional teacher group for each module to provide teaching materials for service sites and personnel empowerment training.

(2) Data collection steps After the stronghold and Rizhao agreed to cooperate with the "Experts' Suggestion on Curriculum Adjustment", the first data collection was carried out, and then the new curriculum adjustment was carried out for three months, and then two data collections were carried out. The researchers conducted at least three to four times on these strongholds and Rizhao data collection (The first complete data collection is completed within one to two weeks before the formal adjustment of the course; the second time is collected within two weeks after the course is implemented for three months; the third time is 6 months after the start of implementation; the fourth time Collected 9-12 months after start of implementation.

(3) Description of the data collection role of the researchers of this project: The objects of data collection are the elders, their families, and caregivers in the bases and Rizhao. The research team only makes suggestions on the courses in the institutions that are willing to participate, and makes suggestions on the implementation of course activities with the personnel who originally booked the courses. It is not the project that sends people to the base or directly leads the activities in Rizhao. The researchers of this project are Facilitator of course activities and data collector or evaluator of effectiveness items.

(4) Objects and contents of data collection in strongholds and Rizhao Data collection content of the elders, their family members, and care workers in the base and Rizhao, except for the data collection content of the first stage In addition, in order to have a more comprehensive understanding of the changes in the performance of the elderly, the functions in the following table 2. will be collected again.

ELIGIBILITY:
Inclusion Criteria:

* Recruit the elders (and their family members) in community bases and Rizhao centers, caregivers of bases and Rizhao centers.

Exclusion Criteria:

* Because the plan hopes to conduct an extensive inventory/detection of the dementia and disability status of the elderly in the dementia stronghold and Rizhao Center, unless the subjects do not want to To join the research, there are no conditions for case scheduling in this plan

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The objects of data collection are the elders, their families, and caregivers in the bases and Rizhao. The research team only makes suggestions on the courses in the institutions that are willing to participate, and makes suggestions on the implementation of course activities with the personnel who originally booked the courses. It is not the project that sends people to the base or directly leads the activities in Rizhao. The researchers of this project are Facilitator of course activities and data collector or evaluator of effectiveness items.
Sampling Method: Non-Probability Sample
Enrollment: 652 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
basic information | Two weeks before intervention
  Including gender, age, height, weight, marital status, education level,
  Gender:
  This pertains to the participant's biological gender and may be identified as either male or female.
  Age:
  Represents the participant's age, typically measured in years.
  Height:
  The participant's height, typically measured in centimeters or inches.
  Weight:
  The participant's weight, typically measured in kilograms or pounds.
  Marital Status:
  Describes the participant's current marital status, such as married, unmarried, divorced, etc.
  Educational Level:
  This indicates the participant's level of education, including degrees or other educational qualifications.
  Medical Conditions:
  Describes the participant's health condition, which may encompass past medical history, current illnesses, or chronic conditions.
cognitive function assessment | Two weeks before intervention
  (SPMSQ - Short Portable Mental Status Questionnaire): Description: SPMSQ, a concise cognitive screening tool, assesses memory and cognitive function via questions on orientation, memory, and mathematical abilities.
  (Mini-Mental State Examination; MMSE): Description: MMSE, widely used for cognitive function assessment, covers domains like orientation, registration, attention, calculation, recall, language, and visuospatial skills.
  (Cognitive Abilities Screening Instrument; CASI): Description: CASI, a comprehensive tool, assesses attention, concentration, orientation, short-term memory, language, and visual construction.
  Scoring: Scores can range from 0 to 100, with higher scores indicating better cognitive function. Specific cutoff scores may be used to identify different levels of cognitive impairment.
Psychiatric and behavioral symptoms | Two weeks before intervention
  Use NPI or other mental behavioral scales that are more suitable for Rizhao elders
  NPI (Neuropsychiatric Inventory):
  Description: The NPI is a tool designed to assess neuropsychiatric behaviors, particularly in the elderly. It covers various domains such as hallucinations, anxiety, depression, insomnia, etc., providing insights into the assessed individual's behavioral symptoms.
  Scoring: Each domain has corresponding scores, and a total score helps assess the severity of neuropsychiatric symptoms.
daily life functions | Two weeks before intervention
  Measured by Pap scale and IADL.
  Barthel Index:
  Description: The Barthel Index assesses an individual's activities of daily living and self-care abilities, especially in rehabilitation and residential care settings. It includes basic activities like eating, bathing, dressing, toileting, etc.
  Scoring: Each activity is assigned specific scores, and the total score is used to evaluate the overall self-care abilities of the individual. Higher scores indicate better daily living skills.
  IADL (Instrumental Activities of Daily Living):
  Description: IADL is used to assess more complex daily living skills, such as shopping, cooking, using the phone, handling finances, etc. These skills reflect an individual's level of independence in social and home settings.
  Scoring: IADL scores are used to evaluate the individual's capabilities in these more complex activities. Higher scores indicate stronger independent abilities.
body movement function | Two weeks before intervention
  Hand Grip Strength:
  Description: Hand grip strength is a test to assess an individual's hand muscle strength, usually measured using a hand dynamometer.
  Single Leg Stand:
  Description: Single leg stand is a test to assess balance and stability, typically requiring the individual to stand on one leg for a certain duration to test their control of the center of gravity.
  Five Times Sit-to-Stand:
  Description: This test assesses lower limb strength and the ability to stand up, requiring the individual to stand up and sit down five times to test muscle strength and coordination.
  Timed Up and Go:
  Description: Timed Up and Go is a test assessing dynamic balance and walking ability. It requires the individual to stand up from a chair, walk a distance, and then return to sit down.
  Walking Speed:
  Description: Walking speed tests assess the individual's speed during walking, serving as an important indicator of daily activity ability and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiun Liaw, Study Director — Kaohsiung Medical University Department of Physical Therapy Associate Professor
Locations (1):
- Lih-Jiun Liaw, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No